CLINICAL TRIAL: NCT06427681
Title: An Open-label, Randomized, Single-dose, Two-period Cross-over Study to Evaluate the Relative Bioavailability Between BH006 for Injection Per the Intended Dosage Regimen and Fosaprepitant and Palonosetron in Healthy Subjects
Brief Title: An Relative Bioavailability Study of BH006 for Injection in Healthy Subjects
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Zhuhai Beihai Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: BH006-BE-102
Record Dates: First submitted 2024-05-08; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Bioavailability
MeSH Terms: interventions — Injections; fosaprepitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BH006 for injection (Experimental): 150 mg fosaprepitant/0.25 mg palonosetron intravenously 30 minutes (±1 minute)
  Interventions: Drug: BH006 for injection
- Fosaprepitant for injection+Palonosetron hydrochloride injection (Active Comparator): Fosaprepitant for injection：150 mg fosaprepitant intravenously 30 minutes (±1 minute) ; Palonosetron hydrochloride injection： 0.25 mg palonosetron in 5 mL (0.05 mg/mL) infusion time is 30 seconds (﹢5seconds) .
  Interventions: Drug: Fosaprepitant for injection+Palonosetron hydrochloride injection

INTERVENTIONS:
Drug: BH006 for injection — According to the random administration plan, the test product BH006 [(fosaprepitant and palonosetron) for injection] 150mg/0.25mg or the reference product [EMEND® (fosaprepitant) for injection 150 mg + Palonosetron hydrochloride injection 0.25 mg) were injected, and crossovered after a sufficient washing period (14 days), dosing is carried out for the second cycle study.
  Arms: BH006 for injection
Drug: Fosaprepitant for injection+Palonosetron hydrochloride injection — According to the random administration plan, the test product BH006 [(fosaprepitant and palonosetron) for injection] 150mg/0.25mg or the reference product [EMEND® (fosaprepitant) for injection 150 mg + Palonosetron hydrochloride injection 0.25 mg) were injected, and crossovered after a sufficient washing period (14 days), dosing is carried out for the second cycle study.
  Other Names: EMEND®+PALONOSETRON
  Arms: Fosaprepitant for injection+Palonosetron hydrochloride injection

SUMMARY:
The study is an open label, randomized, balanced, two period, two sequence, crossover, single dose, relative bioavailability study in healthy subjects.Each subject, meeting all the inclusion criteria and none of the exclusion criteria, will receive test product or reference product in a crossover manner based on randomization schedule. A balance between T-R and R-T randomization sequence will be ensured using statistical techniques. Blood samples for PK assessment will be collected prior to and after start of intravenous infusion on Day 1 (Period I), Day 15 (Period II).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide signed and dated informed consent prior to any study-related procedures.
2. Willing and able to comply with all study procedures.
3. Subjects and their spouses must agree to use adequate contraception 14 days prior to the first dose, for the duration of study participation, and for 6 months following completion of therapy.
4. Healthy subjects of either gender, ≥18 years of age, or ≤ 55 years of age.
5. Have a body weight (BW) of ≥ 45.0 kg(female) / ≥ 50.0 kg(male) and 18 ≤ body mass index (BMI) ≤ 28 kg/m2.
6. Subjects had normal vital signs (T: 35.9~37.6℃; P: 50~100 beats/min; BP: 90~139mmHg/60~89mmHg, all including critical values) and good organ function prior to enrollment:

   * 12-ECG: QTc <450 milliseconds for males and <470 milliseconds for females;
   * Platelets ≥ 100 × 109/L; neutrophil count ≥ 1.5 × 109/L; hemoglobin ≥ 110 g/L;
   * Alanine aminotransferase, aspartate aminotransferase and bilirubin ≤ ULN;
   * Subjects with abnormal values on physical examination and the rest of the laboratory tests were also enrolled if the investigator determined that the abnormality was not clinically significant in the context of past medical history.

Exclusion Criteria:

1. Those who are known to be allergic to the investigational drug, its excipients, or similar drugs, or those who suffer from allergic diseases or belong to an allergic constitution (such as allergies to two or more drugs, food, or pollen).
2. Those who have a history of clinically serious disease and have not been cured, or those who currently have a disease that may significantly affect the PK or safety evaluation of the study drug.
3. Those with abnormal and clinically significant vital signs, 12-ECG, and clinical laboratory tests.
4. Major surgery within 90 days prior to study entry; minor surgery within 2 weeks prior to study entry.
5. Subjects who have received a vaccination within 30 days prior to the first dose.
6. Subjects who have used or using any drug within 30 days prior to the first dose that may have a significant impact on the PK or safety evaluation of this study drug, including, but not limited to, CYP3A4 inhibitors/agonists, drugs that may alter activity of drug metabolizing enzyme of liver.
7. Subjects who have participated in and used any clinical trial drug within 90 days prior to the first dose, or plan to participate in other clinical trials during this study.
8. Those with a history of alcohol abuse, or regular drinkers within 90 days prior to the first dose (14 units of alcohol per week: 1 unit = 285 mL of beer, or 25 mL of spirits, or 100 mL of wine), or those who could not abstain during the test, or had a positive alcohol breath test. (1 unit = 1 unit of alcohol = about 285 mL of beer or about 100 mL of red wine or about 25 mL of beverage containing 40% (v/v) alcohol).
9. Subjects who are addicted to tobacco (more than 5 cigarettes or equivalent per day) within 30 days prior to the first dose, or who were unable to quit smoking during the trial.
10. Subjects who have lost/donated more than 450 mL of blood (except physiological blood loss in females) within 90 days prior to the first dose, or who have received a blood transfusion or used a blood product, or who plan to donate blood during the trial or within 30 days of the end of the trial.
11. Subjects who have taken a special diet (including pitaya, mango, grapefruit, etc.) or have had strenuous exercise, or other factors affecting drug absorption, distribution, metabolism, or excretion within 14 days prior to the first dose.
12. Consumption of food or beverages containing alcoholic products or caffeine or xanthine within 48 hours before the first dose.
13. Subjects have a history of drug abuse within the past five years or a positive drug abuse screen.
14. Subjects have presence of Hepatitis B surface antigen (HBsAg) or a Positive Hepatitis C antibody test result, or positive human immunodeficiency virus (HIV) antibody test, or Positive test for syphilis spirochete antibodies at screening.
15. Female subjects who are pregnant or breastfeeding, or have a positive blood pregnancy test result at screening.
16. Subjects have other clinical significant findings within the 12 months prior to screening that indicate clinically significant disease of the following (including, but not limited to, gastrointestinal, renal, hepatic, neurological, haematological, endocrine, oncological, pulmonary, immunological, psychiatric, or cardiovascular disorders); and suffering from any condition that increases the risk of haemorrhage such as haemorrhoids, acute gastritis, or gastric and duodenal ulcers, intractable constipation.
17. Subjects who have a history of needle sickness, blood sickness or have a problem in collecting blood.
18. Subjects who have an acute illness or concomitant medication from the screening phase until the first dose.
19. Subjects who are engaged in high-altitude work, vehicle driving and other operators of machinery associated with danger.
20. Subjects have other issues that may lead to non-compliance or be unsuitable for inclusion by investigators' judgement.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2024-09 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic Analysis | Period I&Period II：pre-dose to 168.000 hours after starting the infusion.
  The PK endpoints will be studied and assessed by PK parameters for aprepitant and palonosetron:Area Under the Curve From Time 0 Hours to Last Quantifiable Concentration(AUC0-t).
Pharmacokinetic Analysis | Period I&Period II：pre-dose to 168.000 hours after starting the infusion.
  The PK endpoints will be studied and assessed by PK parameters for aprepitant and palonosetron:Area Under the Curve From Time 0 Hours to Infinity(AUC0-∞).
Pharmacokinetic Analysis | Period I&Period II：pre-dose to 168.000 hours after starting the infusion.
  The PK endpoints will be studied and assessed by PK parameters for aprepitant :Maximum Concentration (Cmax).

SECONDARY OUTCOMES:
Pharmacokinetic Analysis | Period I&Period II：pre-dose to 168.000 hours after starting the infusion.
  For aprepitant, aprepitant and palonosetron : Apparent Terminal Elimination Half-Life (t1/2).
Pharmacokinetic Analysis | Period I&Period II：pre-dose to 168.000 hours after starting the infusion.
  For aprepitant, aprepitant and palonosetron : Time to Cmax (Tmax).

OTHER OUTCOMES:
Incidence of Adverse Events [Safety and Tolerability] | from the time of first study drug administration till end of study（ Day24 Visit or Early Termination Visit）
  All adverse events (AE) defined by CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Hong Zhang, PI, Principal Investigator — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No